CLINICAL TRIAL: NCT02812706
Title: A Phase I/II Study of Isatuximab (Anti-CD38 mAb) Administered as a Single Agent in Japanese Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Isatuximab Single Agent Study in Japanese Relapsed AND Refractory Multiple Myeloma Patients
Acronym: Islands
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TED14095; U1111-1175-0679 (Other: UTN)
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1, Cohort 1: Isatuximab 10 mg/kg (Experimental): Participants received Isatuximab 10 milligram per kilogram (mg/kg) intravenous (IV) infusion once every week (QW) for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then every 2 weeks (Q2W) (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable adverse events, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 112 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1, Cohort 2: Isatuximab 20 mg/kg (Experimental): Participants received Isatuximab 20 mg/kg IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then Q2W (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable adverse events, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 137 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2: Isatuximab 20 mg/kg (Experimental): Participants received Isatuximab 20 mg/kg IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then Q2W (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable adverse events, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 248 weeks).
  Interventions: Drug: Isatuximab SAR650984

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: solution Route of administration: intravenous
  Other Names: Sarclisa

SUMMARY:
Primary Objectives:

* Phase I: To evaluate safety and tolerability of isatuximab in Japanese participants with relapsed and refractory multiple myeloma.
* Phase II: To evaluate efficacy of isatuximab at recommended dose and to further evaluate the overall response rate (ORR) of isatuximab in Japanese participants with relapsed and refractory multiple myeloma.

Secondary Objectives:

* To evaluate the safety including immunogenicity of isatuximab. The severity, frequency and incidence of all adverse events were assessed.
* To evaluate the pharmacokinetic (PK) profile of isatuximab in the proposed dosing schedule.
* To assess the efficacy using International Myeloma Working Group (IMWG) uniform response criteria.
* To assess the relationship between Baseline cluster of differentiation 38 (CD38) receptor density on multiple myeloma cells and efficacy.

DETAILED DESCRIPTION:
The study duration for an individual participant included a screening period for inclusion of up to 21 days, the treatment period consisting of 28-day cycles and a follow-up period. Treatment with isatuximab might continue until disease progression, unacceptable adverse event, or other reason for discontinuation.

ELIGIBILITY:
Inclusion criteria:

* Males or females, age 20 years or older.
* Participants had a known diagnosis of symptomatic multiple myeloma.
* Participants had received at least 3 prior lines of therapies OR participants whose disease was double refractory to an Immunomodulatory Drug (IMiD) and a Proteasome Inhibitor (PI).
* Participants had been responsive (i.e., minimal response [MR] or better) to at least one prior line of therapy.
* Refractory to the most recently received IMiD or PI included therapy.
* Participants with measurable disease defined as at least one of the following:
* Immunoglobulin G (IgG) Type: Serum M-protein >=1 gram per deciliter (g/dL) (>=10 g/L);
* Immunoglobulin A (IgA) and D Type: Serum M-protein, quantification should be performed;
* Urine M-protein ≥200 mg/24 hours.
* Participants with a Eastern Cooperative Oncology Group (ECOG) performance status <=2.

Exclusion criteria:

* Participants treated with any anti-CD38 agent.
* Diagnosed or treated for another malignancy within 5 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low-risk prostate cancer after curative therapy.
* Prior anticancer therapy (chemotherapy, targeted agents, immunotherapy) within 21 days prior to the first drug infusion unless otherwise specified below:
* Alkylating agents (e.g., Melphalan) within 28 days prior to the first dose of study treatment.
* Steroids treatment (e.g., prednisone greater than (>)10 mg/day orally or equivalent except patients being treated for adrenal insufficiency/replacement therapy or treated for inhalation corticosteroids) within 14 days prior to the first dose of study treatment.
* Participated in another clinical trial within 30 days prior to the first dose of study treatment.
* Participants treated with systemic radiation therapy within 4 weeks prior to the first dose of study treatment OR Localized radiation therapy within 1 week prior to the first dose of study treatment.
* Major surgical procedure within 4 weeks prior to the first dose of study treatment.
* Any toxicity Grade >=2 (excluding alopecia, neutropenia or neuropathy) related to any prior anti-cancer therapy according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
* Neuropathy Grade >=3 or painful peripheral neuropathy Grade >=2.
* History of significant cardiovascular disease unless the disease within the past 6 months was well-controlled.
* Previously received an allogenic stem cell transplant.
* Diagnosed Crow-Fukase (POEMS) syndrome OR plasma cell leukemia.
* Participants with known or suspected amyloidosis.
* Participants with Waldenstrom's macroglobulinemia OR Multiple myeloma IgM subtype.
* Participants with active infection.
* Known human immunodeficiency virus (HIV) or active hepatitis B or C viral infection.
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation.
* Any severe underlying medical conditions including presence of laboratory abnormalities, which could impair the ability to participate in the study or the interpretation of its results.
* Hypersensitivity or history of intolerance to boron or mannitol, sucrose, histidine (as base and hydrochloride salt) and polysorbate 80 or any of the components of study therapy that are not amenable to pre-medication with steroids and H2 blockers or would prohibit further treatment with these agents.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Japan (13):
  - Investigational Site Number :392001, Nagoya, Aichi-ken
  - Investigational Site Number :392005, Shibukawa-shi, Gunma
  - Investigational Site Number :392010, Hiroshima, Hiroshima
  - Investigational Site Number :392015, Kanazawa, Ishikawa-ken
  - Investigational Site Number :392016, Kyoto, Kyoto
  - Investigational Site Number :392008, Suwa-shi, Nagano
  - Investigational Site Number :392003, Okayama, Okayama-ken
  - Investigational Site Number :392009, Osaka, Osaka
  - Investigational Site Number :392013, Suita-shi, Osaka
  - Investigational Site Number :392017, Sunto-gun, Shizuoka
  - Investigational Site Number :392012, Chuo-ku, Tokyo
  - Investigational Site Number :392002, Shibuya-ku, Tokyo
  - Investigational Site Number :392011, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Sunami K, Fuchida SI, Suzuki K, Ri M, Matsumoto M, Shimazaki C, Asaoku H, Shibayama H, Ishizawa K, Takamatsu H, Ikeda T, Maruyama D, Imada K, Uchiyama M, Kiguchi T, Iyama S, Murakami H, Onishi R, Tada K, Iida S. Anti-CD38 antibody isatuximab monotherapy for Japanese individuals with relapsed/refractory multiple myeloma: An update of the phase 1/2 ISLANDs study. Hematol Oncol. 2023 Aug;41(3):442-452. doi: 10.1002/hon.3105. Epub 2022 Dec 15. PMID 36433829
- [Result] Sunami K, Suzuki K, Ri M, Matsumoto M, Shimazaki C, Asaoku H, Shibayama H, Ishizawa K, Takamatsu H, Ikeda T, Maruyama D, Kaneko H, Uchiyama M, Kiguchi T, Iyama S, Murakami H, Takahashi K, Tada K, Mace S, Guillemin-Paveau H, Iida S. Isatuximab monotherapy in relapsed/refractory multiple myeloma: A Japanese, multicenter, phase 1/2, safety and efficacy study. Cancer Sci. 2020 Dec;111(12):4526-4539. doi: 10.1111/cas.14657. Epub 2020 Oct 15. PMID 32975869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in Japan. A total of 36 participants were enrolled between 05 September 2016 and 6 April 2018, and received isatuximab monotherapy.
Pre-assignment Details: Study consisted of 2 phases: Phase 1 and Phase 2. Phase I (Cohorts 1 and 2) was a dose escalation part to evaluate the safety, pharmacokinetics (PK), and efficacy of isatuximab. Phase 2 was commenced after completion of the DLT observation period in Phase 1 and determination of the recommended dose to be used in Phase 2.
Groups:
- Phase 1, Cohort 1: Isatuximab 10 mg/kg: Participants received Isatuximab 10 milligram per kilogram (mg/kg) intravenous (IV) infusion once every week (QW) for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then every 2 weeks (Q2W) (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable adverse events (AEs), disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 112 weeks).
- Phase 1, Cohort 2: Isatuximab 20 mg/kg: Participants received Isatuximab 20 mg/kg IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then Q2W (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 137 weeks).
- Phase 2: Isatuximab 20 mg/kg: Participants received Isatuximab 20 mg/kg IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then Q2W (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 248 weeks).
Period: Phase 1
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg | Phase 2: Isatuximab 20 mg/kg
Started | 3 | 5 | 0 (Phase 1 and Phase 2 were separate populations.)
Completed | 0 | 0 | 0
Not Completed | 3 | 5 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Progressive disease | 3 | 3 | 0
Period: Phase 2
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg | Phase 2: Isatuximab 20 mg/kg
Started | 0 (Phase 1 and Phase 2 were separate populations) | 0 (Phase 1 and Phase 2 were separate populations.) | 28
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 28
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Progressive disease | 0 | 0 | 22
Not completed — Other-Unspecified | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all treated population which included all participants who gave their informed consent and received at least one dose (even incomplete) of isatuximab.
Groups:
- Phase 1, Cohort 1: Isatuximab 10 mg/kg: Participants received Isatuximab 10 mg/kg IV infusion QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1), and then Q2W (i.e., on Day 1 and 15) for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs, disease progression, or any other reason for discontinuation whichever occurs first (maximum duration of exposure: 112 weeks).
- Total: Total of all reporting groups
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg | Phase 2: Isatuximab 20 mg/kg | Total
Number analyzed (Participants) | 3 | 5 | 28 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.6) | 74.4 (4.7) | 70.6 (8.1) | 70.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 10 | 16
  Male | 1 | 1 | 18 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 28 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs: AEs occurring during 1st treatment cycle, assessed per national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) version 4.03. DLTs included: Hematologic DLTs: Grade(G) 4 neutropenia(N) lasting greater than or equal to (>=) 5 days; G3 to G4 N with fever or microbiologically or radiographically documented infection; G4 thrombocytopenia lasting for >=5 days; thrombocytopenia, treatment delay greater than (>)14 days due to hematologic toxicity. Non-hematologic DLTs: G>=3 non-hematological AE, excluding G3 fatigue, G 3 to 4 electrolyte abnormalities, G3 nausea/vomiting/diarrhea if responsive to optimal medical management within 48 hours or allergic reaction/ hypersensitivity attributed to isatuximab; AE that required treatment delay for >14 days. Any other toxicity deemed by Investigator or sponsor to be dose-limiting, regardless of the grade, was also considered DLT.
Time Frame: Cycle 1 (28 days)
Population: Analysis was performed on DLT evaluable population that included subset of participants who completed the first Cycle which consisted of 4 isatuximab administrations of the study drug or they discontinued study drug before completion of first cycle for a DLT.
  .
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

2. Primary Outcome: Phase 2: Percentage of Participants With Overall Response (OR)
Description: Percentage of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) assessed by International Myeloma Working Group (IMWG) uniform response criteria. sCR: CR as defined plus normal FLC ratio & absence of clonal cells in bone marrow. CR: negative immunofixation on serum & urine; disappearance of any soft tissue plasmacytomas; <5% plasma cells in bone marrow; normal FLC ratio of 0.26-1.65. VGPR: serum & urine M-protein detectable by immunofixation; >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h; >90% decrease in difference between involved & uninvolved FLC levels required. PR: >=50% reduction of serum M-protein & reduction in 24h urinary M protein by >=90%/<200 mg/24 h; if serum & urine M-protein unmeasurable:>=50% decrease in difference between involved & uninvolved FLC; if serum & urine M-protein not measurable:>=50% reduction in plasma cells required, in place of M-protein.
Time Frame: From the date of the first response until the primary analysis data cut-off date of 31 July 2018 (median duration of follow-up was 24.14 weeks)
Population: Analysis was performed on all treated population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
percentage of participants | 32.1

3. Secondary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation patient administered with a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TESAEs was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that develop, worsened or became serious during the on-treatment period (time from first dose of study drug up to 30 days after the last dose of study drug administration).
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug administration (maximum duration of exposure: up to 112 weeks for Cohort 1 and 137 weeks for Cohort 2)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 5
Participants
  TEAEs | 3 | 4
  TESAEs | 1 | 2

4. Secondary Outcome: Phase 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation patient administered with a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. TESAEs was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs are defined as AEs that develop, worsened or became serious during the on-treatment period (time from first dose of study drug up to 30 days after the last dose of study drug administration).
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug administration (maximum duration of exposure: up to 248 weeks)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
Participants
  TEAEs | 25
  TESAEs | 11

5. Secondary Outcome: Phase 1: Percentage of Participants With Overall Response (OR)
Description: Percentage of participants with sCR, CR, VGPR, and PR assessed by IMWG uniform response criteria. sCR: CR as defined plus normal FLC ratio & absence of clonal cells in bone marrow. CR: negative immunofixation on serum & urine; disappearance of any soft tissue plasmacytomas; <5 percentage (%) plasma cells in bone marrow; normal FLC ratio of 0.26-1.65. VGPR: serum & urine M-protein detectable by immunofixation; >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hour (h); >90% decrease in difference between involved & uninvolved FLC levels required. PR: >=50% reduction of serum M-protein & reduction in 24h urinary M protein by >=90%/<200 mg/24 h; if serum & urine M-protein unmeasurable:>=50% decrease in difference between involved & uninvolved FLC; if serum & urine M-protein not measurable:>=50% reduction in plasma cells required, in place of M-protein.
Time Frame: From the date of the first response until disease progression, or death due to any cause, whichever comes first (maximum duration of exposure: up to 112 weeks for Cohort 1 and 137 weeks for Cohort 2)
Population: Analysis was performed on all treated population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 5
percentage of participants | 66.7 | 60.0

6. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR: time (in weeks) from date of first response to date of subsequent progressive disease (PD) or death, whichever happens earlier. In absence of confirmation of subsequent PD or death before cut-off date, DOR was censored at date of last valid assessment performed or date of initiation of new anticancer treatment, whichever was earlier. PD (IMWG criteria): increase (inc.) of >=25% from lowest response value in any one of following: serum M-component (absolute inc.>=0.5 g/dL) and/or; urine M-component (absolute inc.>=200 mg/24h) and/or, in participants without measurable serum & urine M-protein: difference between involved & uninvolved FLC levels (absolute inc. >10 mg/dL); in participants without measurable serum & urine M-protein and without measurable disease by FLC levels, bone marrow plasma cell % (absolute % >=10%); development of new bone lesions or soft tissue plasmacytomas/definite inc. in size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia.
Time Frame: as for outcome 5
Population: Analysis was performed on a subset of participants who had response.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 2 | 3
weeks | 100.64 (7.78) | 113.90 (18.45)

7. Secondary Outcome: Phase 2: Percentage of Participants With Clinical Benefit (CB)
Description: CB defined as percentage of participants with sCR, CR, VGPR, PR or Minor/minimal response (MR) assessed by IMWG criteria. sCR: CR as defined plus normal FLC ratio & absence of clonal cells. CR: negative immunofixation on serum & urine; disappearance of any soft tissue plasmacytomas; <5% plasma cells in bone marrow; normal FLC ratio: 0.26-1.65. VGPR: serum & urine M-protein detectable by immunofixation; >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24h; >90% decrease in difference between involved & uninvolved FLC levels required. PR: >=50% reduction of serum M-protein & reduction in 24h urinary M protein by >=90%/<200 mg/24 h; if serum & urine M-protein unmeasurable:>=50% decrease in difference between involved & uninvolved FLC; if serum & urine M-protein not measurable:>=50% reduction in plasma cells required. MR: >=25% but <=49% reduction of serum M protein and reduction in 24h urine M protein by 50-89%; 25-49% reduction in size of soft tissue plasmacytomas.
Time Frame: From date of first study treatment administration until first documented response, or death due to any cause, whichever comes first (maximum duration of exposure: up to 248 weeks)
Population: Analysis was performed on all treated population. Data for this outcome measure was not planned to be collected and analyzed for Phase 1.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
percentage of participants | 53.6

8. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival was defined as the time interval (in months) from the date of first study treatment administration to death due to any cause. In the absence of the confirmation of death before the cut-off date, OS was censored at the last date the participant was known to be alive or at the study cut-off date, whichever was earlier. Analysis was performed by Kaplan-Meier method.
Time Frame: From date of first study treatment administration to the date of death due to any cause (maximum duration of exposure: up to 248 weeks)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
months | NA [20.24 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to the smaller number of participants with events.

9. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time interval (in months) from date of first study treatment administration until disease progression or death due to any cause, whichever comes first. In absence of PD or death, PFS was censored at date of last valid assessment performed before cut-off date or date of initiation of new anticancer treatment, whichever was earlier. PD (IMWG criteria): inc. of >=25% in any one of following: serum M-component absolute (abs.) inc. >=0.5 g/dL) and/or; urine M-component (abs. inc. >=200 mg/24h) and/or, in participants without measurable serum & urine M-protein, difference between involved & uninvolved FLC levels (abs. inc. >10 mg/dL); in participants without measurable serum & urine M-protein & without measurable disease by FLC levels: bone marrow plasma cell % (abs. % >=10%); definite development of new bone lesions or soft tissue plasmacytomas or definite inc. in size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia.
Time Frame: From date of first study treatment administration until disease progression or death due to any cause, whichever comes first (maximum duration of exposure: up to 248 weeks)
Population: Analysis was performed on all treated population. Analysis was performed by Kaplan-Meier method. Data for this outcome measure was not planned to be collected and analyzed for Phase 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
months | 5.6 [3.75 to 12.98]

10. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as time (in weeks) from date of first response to date of subsequent progressive disease (PD) or death, whichever happens earlier. In absence of confirmation of subsequent PD or death before cut-off date, DOR was censored at date of last valid assessment performed or date of initiation of new anticancer treatment, whichever was earlier. PD (IMWG criteria):inc. of >=25% from lowest response value in any one of following: serum M-component (absolute inc.>=0.5 g/dL) and/or; urine M-component (absolute inc.>=200 mg/24h) and/or, in participants without measurable serum & urine M-protein: difference between involved & uninvolved FLC levels (absolute inc.>10 mg/dL); in participants without measurable serum & urine M-protein and without measurable disease by FLC levels, bone marrow plasma cell % (absolute% >=10%); development of new bone lesions or soft tissue plasmacytomas/definite inc. in size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia.
Time Frame: From the date of first response until disease progression, or death due to any cause, whichever comes first (maximum duration of exposure: up to 248 weeks)
Population: Analysis was performed on a subset of participants who had response.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 9
weeks | 58.70 (29.91)

11. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP: time interval (in months) from date of first study treatment administration to date of first assessed disease progression. In absence of disease progression, TTP was censored at date of last valid assessment performed before cut-off date or date of initiation of new anticancer treatment, whichever was earlier. PD (IMWG criteria): inc. of >=25% from lowest response value in any one of following: serum M-component (absolute inc.>=0.5 g/dL) and/or; urine M-component (absolute inc.>=200 mg/24h) and/or, in participants without measurable serum & urine M-protein: difference between involved & uninvolved FLC levels (absolute inc.>10 mg/dL); in participants without measurable serum & urine M-protein and without measurable disease by FLC levels, bone marrow plasma cell % (absolute% >=10%); development of new bone lesions or soft tissue plasmacytomas/definite inc. in size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia.
Time Frame: From date of first study treatment administration until disease progression, or death due to any cause, whichever comes first (maximum duration of exposure: up to 248 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
months | 5.5 [3.745 to 12.977]

12. Secondary Outcome: Phase 1: Plasma Concentration Observed at the End of Intravenous Infusion (Ceoi) of Isatuximab
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion.
Time Frame: End of infusion on Day 1 of Cycle 1
Population: Analysis was performed on PK population that included all participants who gave their informed consent and received at least one dose (even incomplete) of Isatuximab; with data for at least 1 PK parameter available. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 4
micrograms per milliliter | 122 (21.6) | 246 (51.8)

13. Secondary Outcome: Phase 1: Maximum Observed Concentration (Cmax) After First Infusion of Isatuximab
Description: Cmax was defined as the maximum concentration observed after the first infusion calculated using the non-compartmental analysis.
Time Frame: Cycle 1 Day 1 at 0 hour (pre-dose), mid-infusion (2 hours post-infusion), end of infusion (EOI) and EOI+4-hour, Day 2 (24 hour), Day 3 (48 hour), Day 4 (72 hour) and pre-dose on Day 8 (0 hour)
Population: Analysis was performed on PK population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 4
micrograms per milliliter | 124 (22.9) | 280 (64.4)

14. Secondary Outcome: Phase 1: Time to Reach the Maximum Concentration (Tmax) After First Infusion of Isatuximab
Description: Tmax was defined as the time to reach Cmax, calculated using the non-compartmental analysis after the intravenous infusion.
Time Frame: Cycle 1 Day 1 at 0 hour (pre-dose), mid-infusion (2 hours post-infusion), EOI and EOI+4-hour, Day 2 (24 hour), Day 3 (48 hour), Day 4 (72 hour) and pre-dose on Day 8 (0 hour)
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 4
hours | 2.68 [2.32 to 7.25] | 5.56 [3.28 to 8.48]

15. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Versus Curve Over the Dosing Interval (AUC1-week) After First Infusion of Isatuximab
Description: AUC was defined as area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval.
Time Frame: as for outcome 14
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms*hours per milliliter
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 4
micrograms*hours per milliliter | 9300 (3010) | 21300 (5520)

16. Secondary Outcome: Phase 1: Trough Plasma Concentrations (Ctrough) of Isatuximab
Description: Ctrough was the plasma concentration observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on Cycle 1 Day 8 (C1 D8), C1 D15, C1 D22, C2 D1, C2 D15, C3 D1, C3 D15, C4 D1, C4 D15, C5 D1, C5 D15, C6 D1, C6 D15, C7 D1, C7 D15, C8 D1, C8 D15, C9 D1, C9 D15, C10 D1, C10 D15, C11 D1
Population: Analysis was performed on PK population. Here, "Number analyzed" = participants with available data for each specified category and "0" in the number analyzed field signifies that no participants were available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 5
micrograms per milliliter
  Cycle 1 Day 8 | 23.77 (8.98) | 78.52 (38.49)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 4
  Cycle 1 Day 15 | 71.33 (22.87) | 186.33 (69.29)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 4
  Cycle 1 Day 22 | 124.87 (69.51) | 254.00 (97.45)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 4
  Cycle 2 Day 1 | 135.57 (125.10) | 367.75 (127.45)
  Cycle 2 Day 15: number analyzed (Participants) | 2 | 4
  Cycle 2 Day 15 | 167.80 (154.43) | 419.08 (351.57)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 3 Day 1 | 174.40 (184.70) | 500.98 (426.78)
  Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Cycle 3 Day 15 | 193.50 (154.86) | 347.75 (259.68)
  Cycle 4 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 4 Day 1 | 202.85 (172.75) | 344.30 (286.74)
  Cycle 4 Day 15: number analyzed (Participants) | 2 | 4
  Cycle 4 Day 15 | 184.85 (182.65) | 392.63 (322.70)
  Cycle 5 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 5 Day 1 | 220.40 (228.54) | 608.00 (351.93)
  Cycle 5 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 5 Day 15 | 233.00 (237.59) | 581.33 (356.35)
  Cycle 6 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 6 Day 1 | 267.50 (280.72) | 665.67 (385.34)
  Cycle 6 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 6 Day 15 | 160.60 (116.53) | 714.33 (451.44)
  Cycle 7 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 7 Day 1 | 200.15 (165.25) | 611.67 (342.27)
  Cycle 7 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 7 Day 15 | 254.50 (228.40) | 641.67 (246.78)
  Cycle 8 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 8 Day 1 | 303.00 (278.60) | 874.67 (408.85)
  Cycle 8 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 8 Day 15 | 242.50 (88.39) | 789.67 (525.08)
  Cycle 9 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 9 Day 1 | 269.00 (147.08) | 722.67 (379.50)
  Cycle 9 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 9 Day 15 | 444.00 (463.86) | 758.33 (393.20)
  Cycle 10 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 10 Day 1 | 436.50 (441.94) | 941.67 (576.67)
  Cycle 10 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 10 Day 15 | 684.00 (772.16) | 1224.67 (719.96)
  Cycle 11 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 11 Day 1 | 592.00 |

17. Secondary Outcome: Phase 2: Maximum Observed Concentration (Cmax) After First Infusion of Isatuximab
Description: Cmax was predicted using population pharmacokinetic model.
Time Frame: Multiple timepoints from Cycle 1 to Cycle 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
micrograms per milliliter | 747.83 (743.83)

18. Secondary Outcome: Phase 2: Area Under the Plasma Concentration Versus Curve Over the Dosing Interval (AUC1-Week) After First Infusion of Isatuximab
Description: AUC was predicted using population pharmacokinetic model.
Time Frame: Multiple timepoints from Cycle 1 to Cycle 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms * hours per milliliter
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
micrograms * hours per milliliter | 65071 (55554)

19. Secondary Outcome: Phase 2: Trough Plasma Concentrations (Ctrough) of Isatuximab
Description: Ctrough was the plasma concentration observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on C1 D8, C1 D15, C1 D22, C2 D1, C2 D15, C3 D1, C3 D15, C4 D1, C4 D15, C5 D1, C5 D15, C6 D1, C6 D15, C7 D1, C7 D15, C8 D1, C8 D15, C9 D1, C9 D15, C10 D1, C10 D15
Population: Analysis was performed on PK population. Here, "Number analyzed" = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
micrograms per milliliter
  Cycle 1 Day 8: number analyzed (Participants) | 27
  Cycle 1 Day 8 | 376.34 (666.40)
  Cycle 1 Day 15: number analyzed (Participants) | 26
  Cycle 1 Day 15 | 662.52 (1283.39)
  Cycle 1 Day 22: number analyzed (Participants) | 27
  Cycle 1 Day 22 | 604.17 (996.78)
  Cycle 2 Day 1: number analyzed (Participants) | 24
  Cycle 2 Day 1 | 927.63 (1194.16)
  Cycle 2 Day 15: number analyzed (Participants) | 23
  Cycle 2 Day 15 | 826.15 (958.75)
  Cycle 3 Day 1: number analyzed (Participants) | 24
  Cycle 3 Day 1 | 734.39 (675.85)
  Cycle 3 Day 15: number analyzed (Participants) | 20
  Cycle 3 Day 15 | 689.85 (715.21)
  Cycle 4 Day 1: number analyzed (Participants) | 17
  Cycle 4 Day 1 | 723.76 (802.83)
  Cycle 4 Day 15: number analyzed (Participants) | 17
  Cycle 4 Day 15 | 619.35 (356.21)
  Cycle 5 Day 1: number analyzed (Participants) | 17
  Cycle 5 Day 1 | 647.24 (338.97)
  Cycle 5 Day 15: number analyzed (Participants) | 16
  Cycle 5 Day 15 | 683.90 (391.48)
  Cycle 6 Day 1: number analyzed (Participants) | 15
  Cycle 6 Day 1 | 674.20 (439.78)
  Cycle 6 Day 15: number analyzed (Participants) | 14
  Cycle 6 Day 15 | 742.93 (420.34)
  Cycle 7 Day 1: number analyzed (Participants) | 12
  Cycle 7 Day 1 | 733.83 (373.26)
  Cycle 7 Day 15: number analyzed (Participants) | 11
  Cycle 7 Day 15 | 786.27 (331.38)
  Cycle 8 Day 1: number analyzed (Participants) | 11
  Cycle 8 Day 1 | 870.09 (443.79)
  Cycle 8 Day 15: number analyzed (Participants) | 9
  Cycle 8 Day 15 | 1004.00 (463.82)
  Cycle 9 Day 1: number analyzed (Participants) | 8
  Cycle 9 Day 1 | 946.25 (369.91)
  Cycle 9 Day 15: number analyzed (Participants) | 8
  Cycle 9 Day 15 | 878.63 (313.39)
  Cycle 10 Day 1: number analyzed (Participants) | 8
  Cycle 10 Day 1 | 823.75 (314.95)
  Cycle 10 Day 15: number analyzed (Participants) | 8
  Cycle 10 Day 15 | 845.38 (322.48)

20. Secondary Outcome: Phase 1 and 2: CD38 Receptor Density at Baseline
Description: CD38 receptor density assessed from bone marrow aspirates for responder and non-responders' participants was reported.
Time Frame: At Baseline (Day 1)
Population: Participants treated with Isatuximab (Phase 1 and 2) and evaluable for CD38 receptor density assessment. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: sMEC
Groups:
- Non-responder: Participants treated with Isatuximab, with independent adjudication committee assessment response <PR.
- Responder: Participants treated with Isatuximab, with independent adjudication committee assessment response >=PR.
Arm/Group | Non-responder | Responder
Number analyzed (Participants) | 18 | 14
sMEC | 113226.2 (93628.7) | 133378.2 (55518.5)

21. Secondary Outcome: Phase 1: Number of Participants With Anti-drug Antibodies (ADA) Response Against Isatuximab
Description: ADA were categorized as: treatment induced, and treatment boosted response. Treatment-induced ADA: ADA that developed at any time during the ADA on-study observation period in participants without preexisting ADA (ADA that was present in samples drawn during the ADA pretreatment period). Treatment boosted ADA: Preexisting ADA with an increase in titer value between pretreatment & posttreatment samples of at least two titer steps, during the ADA on-study observation period.
Time Frame: From first dose of study drug up to 30 days after last study drug administration (maximum duration of exposure: up to 112 weeks for Cohort 1, and 137 weeks for Cohort 2)
Population: Analysis was performed on ADA population which included all participants that received isatuximab in Phase 1 part of the study, with at least one ADA assessment reportable during the ADA on-study observation periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 3 | 5
Participants
  Treatment-induced ADA | 0 | 0
  Treatment boosted ADA | 0 | 0

22. Secondary Outcome: Phase 2: Number of Participants With Anti-drug Antibodies (ADA) Response Against Isatuximab
Description: as for outcome 21
Time Frame: From first dose of study drug up to 30 days after last study drug administration (maximum duration of exposure: up to 248 weeks)
Population: Analysis was performed on ADA population which included all participants that received isatuximab in Phase 2 part of the study, with at least one ADA assessment reportable during the ADA on-study observation periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Isatuximab 20 mg/kg
Number analyzed (Participants) | 28
Participants
  Treatment-induced ADA | 6
  Treatment boosted ADA | 0

ADVERSE EVENTS:
Time Frame: AE data was collected from first dose of study drug up to 30 days after last dose of study drug administration (maximum duration of exposure: up to 112 weeks for Cohort 1, and 137 weeks for Cohort 2 for Phase 1 part; and up to 248 weeks for Phase 2 part)
Description: All-Cause Mortality data collected during the study was assessed for all enrolled participants. Serious and Other Adverse Events were collected for safety population only (i.e., all participants who gave their informed consent and received at least one dose [even incomplete] of isatuximab).
Arm/Group | Phase 1, Cohort 1: Isatuximab 10 mg/kg | Phase 1, Cohort 2: Isatuximab 20 mg/kg | Phase 2: Isatuximab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/5 | 10/28
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 11/28
Other Adverse Events (participants affected / at risk) | 3/3 | 4/5 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Cohort 1: Isatuximab 10 mg/kg (N=3) | Phase 1, Cohort 2: Isatuximab 20 mg/kg (N=5) | Phase 2: Isatuximab 20 mg/kg (N=28)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Neurogenic Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Cohort 1: Isatuximab 10 mg/kg (N=3) | Phase 1, Cohort 2: Isatuximab 20 mg/kg (N=5) | Phase 2: Isatuximab 20 mg/kg (N=28)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infected Dermal Cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (6) | 1 (1) | 6 (17)
Pharyngitis (Infections and infestations) | 1 (3) | 0 (0) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 4 (9)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 6 (12)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 12 (13)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02812706/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02812706/SAP_001.pdf